CLINICAL TRIAL: NCT04292769
Title: Clinical Study of Descitabine Enhanced Infusion of Autologous DC-CIK Cells as a Post-remission Treatment for Malignant Tumors
Brief Title: Clinical Study of DC-CIK Cells as a Post-remission Treatment for Malignant Tumors
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li Yu (Other)
Responsible Party: Sponsor-Investigator, Li Yu, Principal Investigator, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ONCO-CIK-001
Record Dates: First submitted 2020-02-24; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Malignant Neoplasm
Keywords: Decitabine; dendritic cell-cytokine induced killer
MeSH Terms: conditions — Neoplasms | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decitabine combined with DC-CIK (Experimental): Test group: decitabine combined with autologous DC-CIK cells infusion: decitabine 10mg / d, intravenous administration of d-5 to d-1, autologous DC-CIK cells infusion: first course: d1-d3 The second course: d14-d16; the total number of cells is about 5-10 × 109; IL-2: 200,000 IU / d subcutaneous injection, the first course: d0-d4, the second course: d13-d17, every 2 weeks 1 course of treatment, 2 courses in total.
  Interventions: Drug: Decitabine; Biological: DC-CIK
- DC-CIK (Active Comparator): Control group: autologous DC-CIK cell infusion: the first course: d1-d3, the second course: d14-d16; the total number of cells is about 5-10 × 109; One course: d0-d4, the second course: d13-d17, 1 course every 2 weeks, a total of 2 courses.
  Interventions: Biological: DC-CIK

INTERVENTIONS:
Drug: Decitabine — Decitabine 10mg / d, intravenous administration d-5 ～ d-1
  Arms: Decitabine combined with DC-CIK
Biological: DC-CIK — Autologous DC-CIK cell infusion: the first course: d1-d3, the second course: d14-d16; the total number of cells is about 5-10 × 109;

SUMMARY:
1. Screening stage
2. Evaluation of disease
3. Grouping of patients
4. Infusion of cells
5. Surveillance of adverse effect

DETAILED DESCRIPTION:
1. Screening stage：All patients must be confirmed by pathology priorily and reachead remission after surgery or chemo- or radiotherapy. All criteria patients must sign informed consent in advance.
2. Evaluation of disease: Systematically assessment of tumor burdern and Physical fitness of all patients.
3. Cell preparation：At least one month after the end of the last chemotherapy, 100ml of peripheral blood was collected, and PBMCs were separated and extracted in the tens of thousands and local hundreds of clean laboratories and DC-CIK cells were prepared.
4. Baseline assessment: Systematically assess various biochemical indicators. Those who do not meet the infusion criteria will withdraw from the study after being confirmed by researchers.
5. Study group: All subjects were randomly divided into test group and control group. The test group was treated with decitabine. The course of treatment was a total of 5 times.
6. Infusion：During cell culture and before transfusion, cells should be subjected to strict quality control tests such as bacteria, fungi, mycoplasma, endotoxin, cell activity, DC and T cell identification, etc. The transfusion can be approved only after the quality control is qualified.
7. Adverse reaction monitoring: DC-CIK infusion was used to closely observe changes in subjects' blood pressure, body temperature, blood routine, blood biochemistry, electrolytes, coagulation, cytokines and organ functions.
8. After the trial is completed, the patient's survival information will be followed up every 3 months by telephone or by visiting the test center.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-70 years (including 18 and 70 years);
2. Pathological and histological examination confirmed a malignant solid tumor;
3. Patients with ECOG score <2, estimated survival time> 3 months.
4. Patients with solid tumors have cleared their lesions after treatment, and are unsuitable or unwilling to receive other anti-tumor treatments such as chemotherapy and radiotherapy;
5. Patients did not receive any anti-cancer treatment such as chemotherapy, radiotherapy, immunotherapy (such as immunosuppressive drugs) within 2-4 weeks before enrollment, and their previous treatment-related toxicities have recovered to <1 (hair loss) , Except for low-level toxicity such as peripheral neuritis);
6. The patient's venous channel is unobstructed, which can meet the needs of intravenous drip;
7. Patients voluntarily participate and sign informed consent, and follow the research treatment plan and visit plan.

Exclusion Criteria:

* 1. Patients use large doses of hormones (except for patients using inhaled hormones) within 1 week before enrollment; 2. People with severe autoimmune diseases, immunodeficiency diseases or severe allergies; 3. Patients treated with other cellular immune products (DC, T, NK, and CAR-T, etc.); 4. Patients have uncontrollable infections within 4 weeks before enrollment; 5. Active HBV DNA> 1000copy / mL / Hepatitis C virus (anti-HCV positive, HCV RNA positive), HIV positive, syphilis positive; 6. Patients participated in other clinical studies within 6 weeks before enrollment; 7. Patients with mental illness; 8. Patients with a substance abuse / addiction and medical, psychological or social conditions that may interfere with the study or influence the evaluation of the study results; 9. Alcohol dependence in patients; 10. Women who are pregnant (positive urine / blood pregnancy study) or breastfeeding; men or women with a pregnancy plan in the past year; patients cannot guarantee effective contraception during the study period 11. At the discretion of the investigator, the patient has other unsuitable conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-01-20 (Estimated); Study Completion 2023-01-20 (Estimated)

PRIMARY OUTCOMES:
OS | up to 2 years
  overall survival rate
PFS | up to 2 years
  progression free survival

SECONDARY OUTCOMES:
objective response rate | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen university general hospital, Shenzhen, China

IPD SHARING:
Plan to Share IPD: No